CLINICAL TRIAL: NCT01130818
Title: Double Blind Placebo Controlled Dose Ranging Study for the Assessment of Safety, Tolerability and Pharmacokinetics of Single Ascending Oral Doses of GLPG0492 in Healthy Subjects and Open Relative Bioavailability Study of Oral Solution Versus Solid Formulation, Fasted and Fed, in Elderly Subjects
Brief Title: First-in-Human Single Ascending Dose of GLPG0492
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: GLPG0492-CL-101
Record Dates: First submitted 2010-05-20; First posted 2010-05-26 (Estimated); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Healthy
Keywords: Safety; Tolerability; Pharmacokinetics; Bioavailability (solid vs solution, fasting vs fed); Young healthy subjects; Elderly healthy subjects
MeSH Terms: interventions — 4-(4-(hydroxymethyl)-3-methyl-2,5-dioxo-4-phenylimidazolidin-1-yl)-2-(trifluoromethyl)benzonitrile

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): single ascending doses
  Interventions: Drug: GLPG0492
- 2 (Placebo Comparator): single dose placebo
  Interventions: Drug: placebo
- 3 (Experimental): single dose, oral solution, 50 mg
  Interventions: Drug: GLPG0492
- 4 (Experimental): single dose, capsules (fasting)
  Interventions: Drug: GLPG0492
- 5 (Experimental): single dose, capsules (fed)
  Interventions: Drug: GLPG0492

INTERVENTIONS:
Drug: GLPG0492 — single ascending doses, oral solution (25 to max. 120 mg/intake, 10 to 200 mg/mL)
  Arms: 1; 3
Drug: placebo — single dose, oral solution
  Arms: 2
Drug: GLPG0492 — single dose, solid formulation, 50 mg (2*25 mg/capsule), fasting
  Arms: 4
Drug: GLPG0492 — single dose, solid formulation, 50 mg (2*25 mg/capsule), after high fat breakfast
  Arms: 5

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of single ascending (SAD) oral dose of GLPG0492 compared to placebo in healthy subjects.

Also, pharmacokinetics (PK) and pharmacodynamics (PD) of GLPG0492 after single oral administration will be evaluated, and, if applicable, the maximum tolerated dose determined. Oral bioavailability (solution vs solid capsule fasting or fed) is evaluated in healthy elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

* healthy male, age 18-50 years (young subjects) OR ≥60 years (elderly subjects)
* BMI between 18-30 kg/m², inclusive
* non-smoker

Exclusion Criteria:

* elevated PSA
* drug or alcohol abuse

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-05; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single ascending doses in healthy young and elderly subjects. | up to 10 days postdose

SECONDARY OUTCOMES:
Pharmacokinetics of single oral doses (solution) in young and elderly subjects. | up to 10 days postdose
Determine oral bioavailability of GLPG0492 given to elderly subjects as oral solution or solid dosage form with or without food. | up to 10 days postdose
Determine the maximum tolerated dose in young subjects. | Up to 10 days postdose

CONTACTS AND LOCATIONS:
Overall Officials: Florence Namour, PhD, Study Director — Galapagos NV; Sofie Mesens, MD, Principal Investigator — SGS Stuivenberg
Locations (1):
- SGS Stuivenberg, Antwerp, Belgium